CLINICAL TRIAL: NCT03698318
Title: Pharmacokinetics Study Assessing Bioavailability of Gingerols and Shogaols After Consumption of Five Ginger Extracts in Healthy Volunteers.
Brief Title: Pharmacokinetics Assessing Bioavailability of Gingerols and Shogaols of Five Ginger Extracts
Acronym: KING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Givaudan France Naturals (Industry)
Collaborators: Biofortis Mérieux NutriSciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-A03645-48
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Healthy Subject
Keywords: Ginger; Pharmacokinetics; Shogaols; Gingerols; Bioavailability
MeSH Terms: interventions — oleoresins; ginger extract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Subject sequence 1 (Experimental): Subject allocation sequence 1. Intervention : the subject will receive the five products (tested product n°1, tested product n°2, tested product n°3, tested product n°4 and tested product n°5) in a certain order of assignment of each study product (which will be randomly attributed to him via the randomization sequence).
  Interventions: Dietary Supplement: Tested product n°1; Dietary Supplement: Tested product n°2; Dietary Supplement: Tested product n°3; Dietary Supplement: Tested product n°4; Dietary Supplement: Tested product n°5
- Subject sequence 2 (Experimental): Subject allocation sequence 2. Intervention : the subject will receive the five products (tested product n°1, tested product n°2, tested product n°3, tested product n°4 and tested product n°5) in a certain order of assignment of each study product (which will be randomly attributed to him via the randomization sequence).
  Interventions: Dietary Supplement: Tested product n°1; Dietary Supplement: Tested product n°2; Dietary Supplement: Tested product n°3; Dietary Supplement: Tested product n°4; Dietary Supplement: Tested product n°5
- Subject sequence 3 (Experimental): Subject allocation sequence 3. Intervention : the subject will receive the five products (tested product n°1, tested product n°2, tested product n°3, tested product n°4 and tested product n°5) in a certain order of assignment of each study product (which will be randomly attributed to him via the randomization sequence).
  Interventions: Dietary Supplement: Tested product n°1; Dietary Supplement: Tested product n°2; Dietary Supplement: Tested product n°3; Dietary Supplement: Tested product n°4; Dietary Supplement: Tested product n°5
- Subject sequence 4 (Experimental): Subject allocation sequence 4. Intervention : the subject will receive the five products (tested product n°1, tested product n°2, tested product n°3, tested product n°4 and tested product n°5) in a certain order of assignment of each study product (which will be randomly attributed to him via the randomization sequence).
  Interventions: Dietary Supplement: Tested product n°1; Dietary Supplement: Tested product n°2; Dietary Supplement: Tested product n°3; Dietary Supplement: Tested product n°4; Dietary Supplement: Tested product n°5
- Subject sequence 5 (Experimental): Subject allocation sequence 5. Intervention : the subject will receive the five products (tested product n°1, tested product n°2, tested product n°3, tested product n°4 and tested product n°5) in a certain order of assignment of each study product (which will be randomly attributed to him via the randomization sequence).
  Interventions: Dietary Supplement: Tested product n°1; Dietary Supplement: Tested product n°2; Dietary Supplement: Tested product n°3; Dietary Supplement: Tested product n°4; Dietary Supplement: Tested product n°5
- Subject sequence 6 (Experimental): Subject allocation sequence 6. Intervention : the subject will receive the five products (tested product n°1, tested product n°2, tested product n°3, tested product n°4 and tested product n°5) in a certain order of assignment of each study product (which will be randomly attributed to him via the randomization sequence).
  Interventions: Dietary Supplement: Tested product n°1; Dietary Supplement: Tested product n°2; Dietary Supplement: Tested product n°3; Dietary Supplement: Tested product n°4; Dietary Supplement: Tested product n°5
- Subject sequence 7 (Experimental): Subject allocation sequence 7. Intervention : the subject will receive the five products (tested product n°1, tested product n°2, tested product n°3, tested product n°4 and tested product n°5) in a certain order of assignment of each study product (which will be randomly attributed to him via the randomization sequence).
  Interventions: Dietary Supplement: Tested product n°1; Dietary Supplement: Tested product n°2; Dietary Supplement: Tested product n°3; Dietary Supplement: Tested product n°4; Dietary Supplement: Tested product n°5
- Subject sequence 8 (Experimental): Subject allocation sequence 8. Intervention : the subject will receive the five products (tested product n°1, tested product n°2, tested product n°3, tested product n°4 and tested product n°5) in a certain order of assignment of each study product (which will be randomly attributed to him via the randomization sequence).
  Interventions: Dietary Supplement: Tested product n°1; Dietary Supplement: Tested product n°2; Dietary Supplement: Tested product n°3; Dietary Supplement: Tested product n°4; Dietary Supplement: Tested product n°5
- Subject sequence 9 (Experimental): Subject allocation sequence 9. Intervention : the subject will receive the five products (tested product n°1, tested product n°2, tested product n°3, tested product n°4 and tested product n°5) in a certain order of assignment of each study product (which will be randomly attributed to him via the randomization sequence).
  Interventions: Dietary Supplement: Tested product n°1; Dietary Supplement: Tested product n°2; Dietary Supplement: Tested product n°3; Dietary Supplement: Tested product n°4; Dietary Supplement: Tested product n°5
- Subject sequence 10 (Experimental): Subject allocation sequence 10. Intervention : the subject will receive the five products (tested product n°1, tested product n°2, tested product n°3, tested product n°4 and tested product n°5) in a certain order of assignment of each study product (which will be randomly attributed to him via the randomization sequence).
  Interventions: Dietary Supplement: Tested product n°1; Dietary Supplement: Tested product n°2; Dietary Supplement: Tested product n°3; Dietary Supplement: Tested product n°4; Dietary Supplement: Tested product n°5

INTERVENTIONS:
Dietary Supplement: Tested product n°1 — 1 capsule (26% of gingerol/shogaol in 100 mg) to consume one time for each subject, at one experimental session (random assignment), with 250 mL of water (consumption at T0 time-point of the kinetic)
  Other Names: Gingest TM 26% 28.9 mg
Dietary Supplement: Tested product n°2 — 1 capsule (38.6% of gingerol/shogaol in 74.9 mg) to consume one time for each subject, at one experimental session (random assignment), with 250 mL of water (consumption at T0 time-point of the kinetic)
  Other Names: Oleoresin 39% 28.9 mg
Dietary Supplement: Tested product n°3 — 2 capsules (6.8% of gingerol/shogaol in 424.3 mg) to consume one time for each subject, at one experimental session (random assignment), with 250 mL of water (consumption at T0 time-point of the kinetic)
  Other Names: Ginger 5% 28.9 mg
Dietary Supplement: Tested product n°4 — 1 capsule (27% of gingerol/shogaol in 104.9 mg) to consume one time for each subject, at one experimental session (random assignment), with 250 mL of water (consumption at T0 time-point of the kinetic)
  Other Names: Gingest TM 26% NOP80 28.9 mg
Dietary Supplement: Tested product n°5 — 6 capsules (1.6% of gingerol/shogaol in 1806.25 mg) to consume one time for each subject, at one experimental session (random assignment), with 250 mL of water (consumption at T0 time-point of the kinetic)
  Other Names: Ginger 1.6% 28.9 mg

SUMMARY:
The objective of this study is to assess bioavailability of total gingeroids, free gingerols and shogaols, so as their glucuronide and sulfate metabolites, in the plasma, after consumption of a single dose of 5 different ginger extracts. These five extracts have the same quantity of active substance but with different titration (1.6%, 5%, 39%, 26% and 26% NOP80).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 55 years (limits included),
* BMI between 18.5 and 25 kg/m² (limits included),
* Weight stable within +/- 5% in the last 3 months,
* For women : non menopausal with the same reliable contraception since at least 3 cycles before the beginning of the study and agreeing to keep it during the entire duration of the study (condom with spermicidal gel and estrogen/progestin combination contraception accepted) or menopausal without or with hormone replacement therapy (estrogenic replacement therapy begun from less than 3 months excluded),
* Non smoking or with tobacco consumption ≤ 5 cigarettes / day and agreeing not to smoke during all experimental sessions (V1 to V5),
* Agreeing not to consume food, drink and condiment containing ginger during the all duration of the study,
* Good general and mental health with in the opinion of the investigator: non clinically significant and relevant abnormalities of medical history or physical examination,
* Able and willing to participate to the study by complying with the protocol procedures as evidenced by his dated and signed informed consent form,
* Affiliated with a social security scheme,
* Agreeing to be registered on the volunteers in biomedical research file.

Exclusion Criteria:

* Suffering from a metabolic or endocrine disorder such as diabetes, uncontrolled or controlled thyroidal trouble or other metabolic disorder,
* Suffering from a severe chornic disease (e.g. cancer, HIV, renal failure, ongoing hepatic or biliary disorders, chronic inflammatory digestive disease, arthritis or other chronic respiratory trouble, etc.) or gastrointestinal disorders found to be inconsistent with the conduct of the study by the investigator (e.g. celiac disease),
* Current disease states that are contraindicated to sujects with dietary supplementation: chronic diarrhea, constipation or abdominal pain, Inflammatory bowel diseases (Crohn's disease or ulcerative colitis), Cirrhosis...,
* Suffering from Irritable Bowel Syndrome (IBS) diagnosed by a medical doctor and treated with chronic medication,
* Suffering from an uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg),
* Having medical history of current pathology which could affect the study results or expose the subject to an additional risk according to the investigator,
* Recent gastroenteritis or food borne illness such as confirmed food poisoning (less than 1 month),
* Who made a blood donation in the 3 months before the V0 visit or intending to make it within 3 months ahead,
* With a low venous capital not allowing to perform kinetic of blood samples according to the investigator's opinion,
* With a known or suspected food allergy or intolerance or hypersensitivity to any of the study products' ingredient and/or of the standard meals,
* Pregnant or lactating women or intending to become pregnant within 3 months ahead,
* On any chronic drug treatment (for example antihypertensive treatment, treatment thyroid, asthma treatment, anxiolytic, antidepressant, lipid-lowering treatment, corticosteroids, phlebotonic, veino-tonic, drug with impact on blood circulation...) excepting oral and local contraceptives,
* Under treatment and/or dietary supplement and/or "health food" which could significantly affect parameters followed during the study according to the investigator (i.e. antibiotics, laxatives, antidiarrheal therapy, containg plant extracts (including ginger extracts), probiotics, prebiotics, symbiotics, vitamins and minerals) or stopped less than 3 months before the V0 visit,
* Regular consumption of food and/or drink and/or condiment containing ginger (gari, pickled ginger, Japanese food, tea or infusion...) defined as at least 3 times per week,
* With significant change in food habits or in physical activity in the 3 months before the V0 visit or not agreeing to keep them unchanged throughout the study,
* With a current or planned in the next 3 months specific diet (hyper or hypocaloric, vegan, vegetarian...) or stopped less than 3 months before the study,
* With a personal history of anorexia nervosa, bulimia or significant eating disorders according to the investigator,
* Consuming more than 3 standard drinks of alcoholic beverage daily for men or 2 daily for women or not agreeing to keep his alcohol consumption habits unchanged throughout the study,
* Having a lifestyle deemed incompatible with the study according to the investigator including high level physical activity (defined as more than 10 hours of significant physical activity a week, walking excluded),
* Taking part in another clinical trial or being in the exclusion period of a previous clinical trial,
* Having received, during the last 12 months, indemnities for clinical trial higher or equal to 4500 Euros,
* Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision,
* Presenting a psychological or linguistic incapability to sign the informed consent,
* Impossible to contact in case of emergency,
* Control record (Glycaemia, GGT, ASAT, ALAT, Urea, Creatinine and Comple Blood Count) with clinically significant abnormality according to the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2018-12-07 (Actual); Study Completion 2018-12-07 (Actual)

PRIMARY OUTCOMES:
AUC of total gingeroids plasmatic concentration | From 0 to 8 hours
  The primary endpoint is the AUC (Area Under the Curve) of total gingeroids (gingerols, shogaols and their metabolites) plasmatic concentration from 0 to 8 hours (AUC0-8h) following consumption of ginger extract (expressed in µg.h/mL) and considering the following time-points: T0 to T480. The primary comparisons are GingestTM 26% 28.9 mg versus Oleroresin 39% 28.9 mg, Gingest TM 26% 28.9 mg versus Ginger 5% 28.9 mg and Gingest TM 26% versus Ginger 1.6% 28.9 mg.

SECONDARY OUTCOMES:
AUC0-8H of total gingeroids plasmatic concentration | From 0 to 8 hours
  AUC of total gingeroids (gingerols, shogaols and their metabolites) plasmatic concentrations from 0 to 8 hours following consumption of each test product (expressed in µg.h/mL) and considering the following time-points : T0 to T480.
  Secondary comparisons are GingestTM 26% NOP80 28.9 mg versus Oleoresin 39% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% 28.9 mg versus GingestTM 26% NOP80 28.9 mg, Ginger 5% 28.9 mg versus Oleoresin 39% 28.9 mg, Ginger 5% 28.9 mg versus Ginger 1.6% 28.9 mg and Oleoresin 39% 28.9 mg versus Ginger 1.6% 28.9 mg
AUC0-8H of each analytes of ginger plasmatic concentration separately | From 0 to 8 hours
  AUC of the analytes (6-, 8-, 10-gingerols; 6-, 8-, 10-gingerols glucuronide; 6-, 8-, 10-gingerols sulfate; 6-, 8-, 10-shogaols; 6-, 8-, 10-shogaols glucuronide and 6-, 8-, 10-shogaols sulfate) plasmatic concentrations from 0 to 8 hours following consumption of each test product (expressed in µg.h/mL) and considering the following time-points : T0 to T480.
  Comparisons of interest are GingestTM 26% 28.9 mg versus Oleroresin 39% 28.9 mg, Gingest TM 26% 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Oleoresin 39% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% 28.9 mg versus GingestTM 26% NOP80 28.9 mg, Ginger 5% 28.9 mg versus Oleoresin 39% 28.9 mg, Ginger 5% 28.9 mg versus Ginger 1.6% 28.9 mg and Oleoresin 39% 28.9 mg versus Ginger 1.6% 28.9 mg
AUC0-24H of each total gingeroids plasmatic concentrations | From 0 to 24 hours
  AUC of total gingeroids (gingerols, shogaols and their metabolites) plasmatic concentrations from 0 to 24 hours following consumption of each test product (expressed in µg.h/mL) and considering the following time-points : T0 to T24H.
  Comparisons of interest are GingestTM 26% 28.9 mg versus Oleroresin 39% 28.9 mg, Gingest TM 26% 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Oleoresin 39% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% 28.9 mg versus GingestTM 26% NOP80 28.9 mg, Ginger 5% 28.9 mg versus Oleoresin 39% 28.9 mg, Ginger 5% 28.9 mg versus Ginger 1.6% 28.9 mg and Oleoresin 39% 28.9 mg versus Ginger 1.6% 28.9 mg
AUC0-24H of each analytes of ginger plasmatic concentration separately | From 0 to 24 hours
  AUC of the analytes (6-, 8-, 10-gingerols; 6-, 8-, 10-gingerols glucuronide; 6-, 8-, 10-gingerols sulfate; 6-, 8-, 10-shogaols; 6-, 8-, 10-shogaols glucuronide and 6-, 8-, 10-shogaols sulfate) plasmatic concentrations from 0 to 24 hours following consumption of each test product (expressed in µg.h/mL) and considering the following time-points : T0 to T24H.
  Comparisons of interest are GingestTM 26% 28.9 mg versus Oleroresin 39% 28.9 mg, Gingest TM 26% 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Oleoresin 39% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% 28.9 mg versus GingestTM 26% NOP80 28.9 mg, Ginger 5% 28.9 mg versus Oleoresin 39% 28.9 mg, Ginger 5% 28.9 mg versus Ginger 1.6% 28.9 mg and Oleoresin 39% 28.9 mg versus Ginger 1.6% 28.9 mg
AUC0-∞ of each analytes of ginger plasmatic concentration separately | From 0 to infinity
  AUC of the analytes (6-, 8-, 10-gingerols; 6-, 8-, 10-gingerols glucuronide; 6-, 8-, 10-gingerols sulfate; 6-, 8-, 10-shogaols; 6-, 8-, 10-shogaols glucuronide and 6-, 8-, 10-shogaols sulfate) plasmatic concentrations from 0 to infinity following consumption of each test product (expressed in µg.h/mL) and considering the following time-points : T0 to T24H.
  Comparisons of interest are GingestTM 26% 28.9 mg versus Oleroresin 39% 28.9 mg, Gingest TM 26% 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Oleoresin 39% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% 28.9 mg versus GingestTM 26% NOP80 28.9 mg, Ginger 5% 28.9 mg versus Oleoresin 39% 28.9 mg, Ginger 5% 28.9 mg versus Ginger 1.6% 28.9 mg and Oleoresin 39% 28.9 mg versus Ginger 1.6% 28.9 mg
AUC0-∞ of total gingeroids plasmatic concentrations | From 0 to infinity
  AUC of total gingeroids (gingerols, shogaols and their metabolites) plasmatic concentrations from 0 to infinity following consumption of each test product (expressed in µg.h/mL) and considering the following time-points : T0 to T24H.
  Comparisons of interest are GingestTM 26% 28.9 mg versus Oleroresin 39% 28.9 mg, Gingest TM 26% 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Oleoresin 39% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% 28.9 mg versus GingestTM 26% NOP80 28.9 mg, Ginger 5% 28.9 mg versus Oleoresin 39% 28.9 mg, Ginger 5% 28.9 mg versus Ginger 1.6% 28.9 mg and Oleoresin 39% 28.9 mg versus Ginger 1.6% 28.9 mg
Half-life time of total gingeroids plasmatic concentrations | 24 hours
  Half-life time of total gingeroids (gingerols, shogaols and their metabolites) plasmatic concentrations following consumption of each test product (expressed in minutes).
  Comparisons of interest are GingestTM 26% 28.9 mg versus Oleroresin 39% 28.9 mg, Gingest TM 26% 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Oleoresin 39% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% 28.9 mg versus GingestTM 26% NOP80 28.9 mg, Ginger 5% 28.9 mg versus Oleoresin 39% 28.9 mg, Ginger 5% 28.9 mg versus Ginger 1.6% 28.9 mg and Oleoresin 39% 28.9 mg versus Ginger 1.6% 28.9 mg
Half-life time of each analytes of ginger plasmatic concentration separately | 24 hours
  Half-life time of the analytes (6-, 8-, 10-gingerols; 6-, 8-, 10-gingerols glucuronide; 6-, 8-, 10- gingerols sulfate; 6-, 8-, 10-shogaols; 6-, 8-, 10-shogaols glucuronide and 6-, 8-, 10-shogaols sulfate plasmatic concentrations following consumption of each test product (expressed in minutes).
  Comparisons of interest are GingestTM 26% 28.9 mg versus Oleroresin 39% 28.9 mg, Gingest TM 26% 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Oleoresin 39% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% 28.9 mg versus GingestTM 26% NOP80 28.9 mg, Ginger 5% 28.9 mg versus Oleoresin 39% 28.9 mg, Ginger 5% 28.9 mg versus Ginger 1.6% 28.9 mg and Oleoresin 39% 28.9 mg versus Ginger 1.6% 28.9 mg
Terminal elimination rate constant of each analytes of ginger plasmatic concentration separately | 24 hours
  Terminal elimination rate constant of the analytes (6-, 8-, 10-gingerols; 6-, 8-, 10-gingerols glucuronide; 6-, 8-, 10- gingerols sulfate; 6-, 8-, 10-shogaols; 6-, 8-, 10-shogaols glucuronide and 6-, 8-, 10-shogaols sulfate) plasmatic concentrations following consumption of each test product.
  Comparisons of interest are GingestTM 26% 28.9 mg versus Oleroresin 39% 28.9 mg, Gingest TM 26% 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Oleoresin 39% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% 28.9 mg versus GingestTM 26% NOP80 28.9 mg, Ginger 5% 28.9 mg versus Oleoresin 39% 28.9 mg, Ginger 5% 28.9 mg versus Ginger 1.6% 28.9 mg and Oleoresin 39% 28.9 mg versus Ginger 1.6% 28.9 mg
Terminal elimination rate constant of total gingeroids plasmatic concentrations | 24 hours
  Terminal elimination rate constant of total gingeroids (gingerols, shogaols and their metabolites) plasmatic concentrations following consumption of each test product.
  Comparisons of interest are GingestTM 26% 28.9 mg versus Oleroresin 39% 28.9 mg, Gingest TM 26% 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Oleoresin 39% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% 28.9 mg versus GingestTM 26% NOP80 28.9 mg, Ginger 5% 28.9 mg versus Oleoresin 39% 28.9 mg, Ginger 5% 28.9 mg versus Ginger 1.6% 28.9 mg and Oleoresin 39% 28.9 mg versus Ginger 1.6% 28.9 mg
Time to peak of total gingeroids plasmatic concentrations | 24 hours
  Time to peak of total gingeroids (gingerols, shogaols and their metabolites) plasmatic concentrations following consumption of each test product (expressed in minutes).
  Comparisons of interest are GingestTM 26% 28.9 mg versus Oleroresin 39% 28.9 mg, Gingest TM 26% 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Oleoresin 39% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% 28.9 mg versus GingestTM 26% NOP80 28.9 mg, Ginger 5% 28.9 mg versus Oleoresin 39% 28.9 mg, Ginger 5% 28.9 mg versus Ginger 1.6% 28.9 mg and Oleoresin 39% 28.9 mg versus Ginger 1.6% 28.9 mg
Time to peak of each analytes of ginger plasmatic concentration | 24 hours
  Time to peak of the analytes (6-, 8-, 10-gingerols; 6-, 8-, 10-gingerols glucuronide; 6-, 8-, 10-gingerols sulfate; 6-, 8-, 10-shogaols; 6-, 8-, 10-shogaols glucuronide and 6-, 8-, 10-shogaols sulfate) plasmatic concentrations following consumption of each test product (expressed in minutes).
  Comparisons of interest are GingestTM 26% 28.9 mg versus Oleroresin 39% 28.9 mg, Gingest TM 26% 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Oleoresin 39% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% 28.9 mg versus GingestTM 26% NOP80 28.9 mg, Ginger 5% 28.9 mg versus Oleoresin 39% 28.9 mg, Ginger 5% 28.9 mg versus Ginger 1.6% 28.9 mg and Oleoresin 39% 28.9 mg versus Ginger 1.6% 28.9 mg
Peak of each analytes of ginger plasmatic concentration | 24 hours
  Peak of the analytes (6-, 8-, 10-gingerols; 6-, 8-, 10-gingerols glucuronide; 6-, 8-, 10-gingerols sulfate; 6-, 8-, 10-shogaols; 6-, 8-, 10-shogaols glucuronide and 6-, 8-, 10-shogaols sulfate) plasmatic concentrations following consumption of each test product (expressed in µg/mL).
  Comparisons of interest are GingestTM 26% 28.9 mg versus Oleroresin 39% 28.9 mg, Gingest TM 26% 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Oleoresin 39% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% 28.9 mg versus GingestTM 26% NOP80 28.9 mg, Ginger 5% 28.9 mg versus Oleoresin 39% 28.9 mg, Ginger 5% 28.9 mg versus Ginger 1.6% 28.9 mg and Oleoresin 39% 28.9 mg versus Ginger 1.6% 28.9 mg
Peak of total gingeroids plasmatic concentrations | 24 hours
  Peak of total gingeroids (gingerols, shogaols and their metabolites) plasmatic concentrations following consumption of each test product (expressed in µg/mL).
  Comparisons of interest are GingestTM 26% 28.9 mg versus Oleroresin 39% 28.9 mg, Gingest TM 26% 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Oleoresin 39% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 1.6% 28.9 mg, GingestTM 26% NOP80 28.9 mg versus Ginger 5% 28.9 mg, Gingest TM 26% 28.9 mg versus GingestTM 26% NOP80 28.9 mg, Ginger 5% 28.9 mg versus Oleoresin 39% 28.9 mg, Ginger 5% 28.9 mg versus Ginger 1.6% 28.9 mg and Oleoresin 39% 28.9 mg versus Ginger 1.6% 28.9 mg

CONTACTS AND LOCATIONS:
Overall Officials: Romain Le Cozannet, PhD, Study Director — Givaudan France Naturals
Locations (1):
- Biofortis Mérieux Nutrisciences, Saint-Herblain, France